CLINICAL TRIAL: NCT03550534
Title: The Effectiveness and Safety of Calcium Carbonate in Chronic Kidney Disease With Normophosphatemia: A Double Blind, Randomized Controlled Trial
Brief Title: The Effectiveness and Safety of Calcium Carbonate in Chronic Kidney Disease With Normophosphatemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Collaborators: Dr Cipto Mangunkusumo General Hospital (Other)
Responsible Party: Principal Investigator, Pringgodigdo Nugroho, MD, Head of Dialysis Unit, Dr Cipto Mangunkusumo General Hospital, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 198/UN2.F1/ETIK/2015
Record Dates: First submitted 2018-05-22; First posted 2018-06-08 (Actual); Last update posted 2018-06-08 (Actual); Status verified 2018-06

CONDITIONS: Chronic Kidney Diseases
Keywords: Calcium carbonate; Chronic kidney disease; Normophosphatemia; FGF23; Phosphate binder
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Calcium Carbonate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Calcium Carbonate (Experimental): Calcium carbonate 3 x 500 mg was given to 23 study participants for 12 weeks
  Interventions: Drug: Calcium Carbonate
- Placebo oral capsule (Placebo Comparator): Placebo oral capsule 3 x 1 was given to 23 study participants for 12 weeks
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Calcium Carbonate — Calcium carbonate was obtained from Pharmacy Department, Faculty of Medicine, University of Indonesia. Subjects were randomized to receive calcium carbonate or placebo for 12 weeks.
  Arms: Calcium Carbonate
Drug: Placebo oral capsule — Placebo oral capsule was also obtained from Pharmacy Department, Faculty of Medicine, University of Indonesia. Subjects were randomized to receive calcium carbonate or placebo for 12 weeks.
  Arms: Placebo oral capsule

SUMMARY:
Background: Patient with stage 3 or 4 chronic kidney disease (CKD) usually has normal level of serum phosphate, due to increased serum fibroblast growth factor-23 (FGF23) level that resulted in increased phosphate urine excretion. On the other hand, serum FGF23 elevation was related to CKD progression, vascular calcification, cardiomegaly, and mortality. This double blind, randomized controlled trial study was conducted to evaluate effectiveness and safety of calcium carbonate administration in stage 3 or 4 CKD patients with normophosphatemia.

Hypothesis: Calcium carbonate administration is effective and safe in chronic kidney disease (CKD) with normophosphatemia.

DETAILED DESCRIPTION:
Cardiovascular disease is the most cause of mortality of chronic kidney disease (CKD) patients. As CKD progresses, the prevalence of cardiovascular disease also increased. Beside traditional cardiovascular risk factor that the investigators have known, some non-traditional cardiovascular risk factors were reported to be associated with cardiovascular disease in CKD patients, which one of them was increased level of fibroblast growth factor-23 (FGF23).[1,2]

FGF23 reduces production of 1,25-vitamin D3 and expression of sodium-phosphate cotransport, and also excretes phosphate through urine. In healthy and CKD population, increased phosphate level resulted in increased production of FGF23. Normophosphatemia state in early to moderate stage of CKD was reported due to body compensation by increasing the level of FGF23. On the other hand, increased serum FGF23 level was related to CKD progression, cardiomegaly, vascular calcification, and mortality.[1] There are several ways to prevent hyperphosphatemia, such as low phosphor intake, phosphate binder administration, and adequate dialysis.[3]

Phosphate binder was reported to give positive effects in CKD patients with hyperphosphatemia. Studies which investigated the use of phosphate binder in CKD patients with normophosphatemia to decrease FGF23 were still limited and the result was controversial.[1]

Therefore, this double blind, randomized controlled trial study investigated the effectiveness and safety of calcium carbonate in early to moderate CKD patients with normophosphatemia in lowering FGF23 levels. Study participant were randomized to receive calcium carbonate or placebo for 12 weeks. Before and after intervention, blood and urine sample were taken to examine serum FGF23, serum phosphate, urine phosphate, ionized calcium, serum calcium, urea, creatinine, estimated glomerular filtration rate (eGFR), and albumin. Effectiveness of calcium carbonate administration was indicated by serum FGF23, while safety was indicated by serum calcium.

ELIGIBILITY:
Inclusion Criteria:

* Stage 3 or 4 chronic kidney disease patient that visit nephrology or endocrinology outpatient clinic of dr. Cipto Mangunkusumo Hospital
* Normal level of serum phosphate
* Agreed to join in this study

Exclusion Criteria:

* Subjects with BMI < 18.5 kg/m2 or > 30 kg/m2
* Consume drugs which may interfere bone mineral metabolism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2015-11-06 (Actual); Primary Completion 2016-12-11 (Actual); Study Completion 2016-12-11 (Actual)

PRIMARY OUTCOMES:
Serum Fibroblast Growth Factor 23 (FGF-23) | 12 weeks
  Serum FGF23 (pg/ml) as cardiovascular risk factor in chronic kidney disease (CKD) was measured and compared between 2 groups before and after intervention

SECONDARY OUTCOMES:
Serum Calcium Level | 12 weeks
  Serum calcium level (mg/dl) was measured and compared between 2 groups before and after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Pringgodigdo Nugroho, MD, Principal Investigator — Indonesia University; Maruhum Bonar H. Marbun, MD, Principal Investigator — Indonesia University; Bella Yunita, MD, Principal Investigator — Indonesia University; Cindy Astrella, MD, BMedSci, Principal Investigator — Indonesia University
Locations (1):
- dr. Cipto Mangunkusumo Hospital, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Isakova T, Xie H, Yang W, Xie D, Anderson AH, Scialla J, Wahl P, Gutierrez OM, Steigerwalt S, He J, Schwartz S, Lo J, Ojo A, Sondheimer J, Hsu CY, Lash J, Leonard M, Kusek JW, Feldman HI, Wolf M; Chronic Renal Insufficiency Cohort (CRIC) Study Group. Fibroblast growth factor 23 and risks of mortality and end-stage renal disease in patients with chronic kidney disease. JAMA. 2011 Jun 15;305(23):2432-9. doi: 10.1001/jama.2011.826. PMID 21673295
- [Result] Martin K, Floege J, Ketteler M. Bone and mineral metabolism in chronic kidney disease. In: Johnson R, Feehally J, Floege J, editors. Comprehensive clinical nephrology. Fifth edition. Philadelphia: Saunders; 2015. p. 984-7.
- [Result] Ketteler M, Leonard M. KDIGO 2016 Clinical practice guideline update on diagnosis, evaluation, prevention, and treatment of CKD-MBD. Off J Int Soc Nephrol. 2016;(August):1-45
- [Result] Prakash S, O'Hare AM. Interaction of aging and chronic kidney disease. Semin Nephrol. 2009 Sep;29(5):497-503. doi: 10.1016/j.semnephrol.2009.06.006. PMID 19751895
- [Result] Iseki K. Gender differences in chronic kidney disease. Kidney Int. 2008 Aug;74(4):415-7. doi: 10.1038/ki.2008.261. PMID 18670407
- [Result] Perhimpunan Nefrologi Indonesia. 8th Report of Indonesian Renal Registry. Jakarta; 2015
- [Result] Bayliss G, Weinrauch LA, D'Elia JA. Pathophysiology of obesity-related renal dysfunction contributes to diabetic nephropathy. Curr Diab Rep. 2012 Aug;12(4):440-6. doi: 10.1007/s11892-012-0288-1. PMID 22638939
- [Result] Langman CB, Cannata-Andia JB. Calcium in chronic kidney disease: myths and realities. Introduction. Clin J Am Soc Nephrol. 2010 Jan;5 Suppl 1:S1-2. doi: 10.2215/CJN.06140809. No abstract available. PMID 20089497
- [Result] Fliser D, Kollerits B, Neyer U, Ankerst DP, Lhotta K, Lingenhel A, Ritz E, Kronenberg F; MMKD Study Group; Kuen E, Konig P, Kraatz G, Mann JF, Muller GA, Kohler H, Riegler P. Fibroblast growth factor 23 (FGF23) predicts progression of chronic kidney disease: the Mild to Moderate Kidney Disease (MMKD) Study. J Am Soc Nephrol. 2007 Sep;18(9):2600-8. doi: 10.1681/ASN.2006080936. Epub 2007 Jul 26. PMID 17656479
- [Result] Soriano S, Ojeda R, Rodriguez M, Almaden Y, Rodriguez M, Martin-Malo A, Aljama P. The effect of phosphate binders, calcium and lanthanum carbonate on FGF23 levels in chronic kidney disease patients. Clin Nephrol. 2013 Jul;80(1):17-22. doi: 10.5414/CN107764. PMID 23391319
- [Result] Shigematsu T, Negi S; COLC Research Group. Combined therapy with lanthanum carbonate and calcium carbonate for hyperphosphatemia decreases serum FGF-23 level independently of calcium and PTH (COLC Study). Nephrol Dial Transplant. 2012 Mar;27(3):1050-4. doi: 10.1093/ndt/gfr388. Epub 2011 Jul 19. PMID 21771755
- [Result] Oliveira RB, Cancela AL, Graciolli FG, Dos Reis LM, Draibe SA, Cuppari L, Carvalho AB, Jorgetti V, Canziani ME, Moyses RM. Early control of PTH and FGF23 in normophosphatemic CKD patients: a new target in CKD-MBD therapy? Clin J Am Soc Nephrol. 2010 Feb;5(2):286-91. doi: 10.2215/CJN.05420709. Epub 2009 Nov 12. PMID 19965540
- [Result] Block GA, Wheeler DC, Persky MS, Kestenbaum B, Ketteler M, Spiegel DM, Allison MA, Asplin J, Smits G, Hoofnagle AN, Kooienga L, Thadhani R, Mannstadt M, Wolf M, Chertow GM. Effects of phosphate binders in moderate CKD. J Am Soc Nephrol. 2012 Aug;23(8):1407-15. doi: 10.1681/ASN.2012030223. Epub 2012 Jul 19. PMID 22822075
- [Result] Sprague SM, Abboud H, Qiu P, Dauphin M, Zhang P, Finn W. Lanthanum carbonate reduces phosphorus burden in patients with CKD stages 3 and 4: a randomized trial. Clin J Am Soc Nephrol. 2009 Jan;4(1):178-85. doi: 10.2215/CJN.02830608. Epub 2008 Dec 3. PMID 19056618
- [Result] Hill KM, Martin BR, Wastney ME, McCabe GP, Moe SM, Weaver CM, Peacock M. Oral calcium carbonate affects calcium but not phosphorus balance in stage 3-4 chronic kidney disease. Kidney Int. 2013 May;83(5):959-66. doi: 10.1038/ki.2012.403. Epub 2012 Dec 19. PMID 23254903